CLINICAL TRIAL: NCT06805838
Title: Prolonged Manual Ventilation Simulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: SafeBVM (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DoD Ventilation Study; HT94252310316 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Manual Ventilation
Keywords: Prolonged manual ventilation simulation; BVM; Sotair; BLS certification; tidal volume; peak inspiratory pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Ambu + Normal lung compliance (No Intervention): Manual ventilation with Ambu bag and normal lung compliance.
- Ambu + Low lung compliance (No Intervention): Manual ventilation with Ambu bag and low lung compliance.
- Smart bag + Normal lung compliance (No Intervention): Manual ventilation with smart bag and normal lung compliance.
- Smart bag + Low lung compliance (No Intervention): Manual ventilation with smart bag and low lung compliance.
- Ambu + Sotair + Normal lung compliance (Active Comparator): Manual ventilation with Ambu bag and Sotair device with normal lung compliance.
  Interventions: Device: Sotair
- Ambu + Sotair + Low compliance (Active Comparator): Manual ventilation with Ambu bag and Sotair device with low lung compliance.
  Interventions: Device: Sotair

INTERVENTIONS:
Device: Sotair — The device is a durable plastic connector with a silicone flap inside it requiring no special handling. There are no patients involved, only a simulated lung that also requires no special handling. Adult Sotair® device has FDA clearance as a Class II device through the 510(k) pathway (K212905) for the intended use of "Flow-limiting, safe, and optimal manual ventilation to minimize gastric insufflation."
  Arms: Ambu + Sotair + Low compliance; Ambu + Sotair + Normal lung compliance

SUMMARY:
A pilot study on simulated lung scenarios using the standard manual resuscitator bag, flow limiting resuscitator bag, and an FDA approved flow rate limiting device paired with a standard manual resuscitator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Have a current basic life support (BLS) certification
* Be available for the entire 10 hours to complete the protocol

Exclusion Criteria:

* Any training in medical school or respiratory therapy school
* Not being available for the full 10 hours to complete the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Minute ventilation while manually ventilating the simulated lung | 10 hours of manual ventilation
  The primary Ventilation endpoint is minute ventilation while manually ventilating the simulated lung over the course of 10 hours.
Minute ventilation while manually ventilating the simulated lung | 10 hours of manual ventilation
  The major endpoints of the subjects response to performing the manual ventilation will be: Respiratory rate and heart rate; Samn-Perelli 7-point fatigue scale reported hourly; Modified Borg Rating of Perceived Exertion 10-point scale reported hourly.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 10 hours of manual ventilation
  Secondary endpoints include: tidal volume, peak inspiratory pressure, respiratory rate, and estimated alveolar ventilation while ventilating the simulated lung.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Brady, MD, Principal Investigator — Brown Physicians, Inc.
Locations (1):
- Brown Physicians, Inc, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
Decision has not been determined.